CLINICAL TRIAL: NCT07340372
Title: Home Monitoring in eAMD Treatment
Acronym: HOME
Status: Not yet recruiting | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2024-15
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Exudative Age-Related Macular Degeneration
Keywords: Aflibercept 8 mg; Exudative Age-Related Macular Degeneration; Patient reported outcomes; Value-based Healthcare; Home monitoring app
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Aflibercept 8mg — Patients will be treated with Aflibercept 8 mg, according to the standard clinical practice, in a treat and extent regimen with the inclusion of a home monitoring application.

SUMMARY:
The goal of this observational clinical study is to collect more information about the efficacy of Aflibercept 8 mg injections in people with eAMD. The main questions it aims to answer are:

* To reassure patients and doctors with longer intervals using home monitoring app;
* To assess patient reported outcomes (PROMs) and Value-based Healthcare.

Participants already taking Aflibercept 8 mg as part of their regular medical care for eAMD will undergo regular ophthalmological examination and use a home monitoring app, in a one year and a two-year treatment period.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) constitutes a degenerative disease of the retina, and it is a major cause of retinal disease in the western world and one of the most common causes of central vision impairment, with the advanced form affecting 1-3% of its total population. Patients with AMD have a reduction in quality of life, as several activities of daily routine require functional central visual perception, such as driving and reading. Population aging will lead to a considerable increase in AMD prevalence. Today, late-stage AMD is the leading cause of blindness among the elderly in industrialized countries and affects more than 2.5 million patients in the European Union (EU) resulting in direct annual costs of over 2 billion Euros.

Advanced forms of AMD (intermediate AMD or late AMD) are seen primarily in 2 types, exudative AMD involving the presence of choroidal neovascularization and nonexudative or dry AMD with geographic atrophy.

Vascular endothelial growth factor (VEGF) is a major pathogenic factor in eAMD and is a signalling protein that is known to be involved in the pathophysiology of angiogenesis and increases vascular permeability. Medical treatment of neovascular (or exudative) AMD (eAMD) has improved considerably due to the introduction of vascular endothelial growth factor inhibitors (anti-VEGF), which have significantly altered the prognosis of the disease.

The current gold standard treatment of eAMD is regular intravitreal injections of anti-VEGF, such as Aflibercept, in a treat-and-extend (T&E) or a fixed regimen. Aflibercept acts as a soluble protein for VEGF receptors inhibiting the predominant signaling pathway responsible for angiogenesis and vascular leakage. Currently, medications like Aflibercept 8 mg are used to treat and manage neovascular age-related macular degeneration, diabetic macular edema, myopic choroidal neovascularization, macular edema associated with retinal vein occlusion, and diabetic retinopathy. However, several patients do not respond adequately to this treatment or suffer a loss of efficacy after multiple administrations. In addition, current treatment with intravitreal anti-VEGF agents is associated with a significant treatment burden and costs for patients, caregivers, and physicians.

With these therapies, longer intervals up to 20 or 24 weeks can be achieved. However, there is a need to have real time information from these patients during such longer intervals, avoiding potential functional and/ or anatomical decline or treatment dropouts. Moreover, it is also pivotal to evaluate potential longer treatment intervals without lower clinical outcomes to reassure the confidence in these longer intervals.

The purpose of home-monitoring is to reduce any delay in the treatment of eAMD. This is through 3 mechanisms:

1. Improved patient literacy: patients being provided with standardised information that helps them to self-care: understanding their disease, treatments and what support services are available, and what the red-flag symptoms are that the patient should be quickly re-presenting to their eye clinic if they encounter.
2. Patient participation in monitoring: remote vision data gathered frequently and viewed by the patient gives them the opportunity for identifying smaller changes at an earlier stage.
3. Clinical teams having access to remote-monitoring vision data: remote vision data gathered frequently and viewed by a specialist gives them the opportunity for identifying smaller changes at an earlier stage, especially with the support of AI-driven algorithms.

Additionally, by helping eAMD patients achieve the best clinical outcomes without the demands of monthly or frequent visits, these new technologies may enhance their quality of life and decrease economic and social burden.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 55 years old) with exudative AMD in the study eye.
* Treatment-naïve patients or patients who have started treatment with IVT anti-VEGF (aflibercept 2 mg, aflibercept 8 mg, faricimab, ranibizumab, bevacizumab, brolucizumab, pegaptanib sodium) up to 48 weeks before inclusion.
* BCVA early treatment diabetic retinopathy study (ETDRS) letter score of 85 to 34 (approximate Snellen equivalent of 20/20 to 20/200) in the study eye with decreased vision determined to be primarily the result of eAMD.
* Willing and able to comply with clinic visits and study-related procedures.
* Provide informed consent signed by study participant or legally acceptable representative.
* Own a working smartphone or tablet compatible with the OKKO Health application.
* Be able to operate the application after training according to OKKO Health indications of use: be alert and mentally competent, has competent dexterity and has normal or corrected hearing to normal audio level.

Exclusion Criteria:

* Evidence of macular edema due to any cause other than eAMD in either eye.
* Other ocular disease in the study eye that could prevent an accurate evaluation of treatment efficacy like, diabetic macular edema, posterior uveitis, corneal opacity, vein occlusion, macular dystrophy.
* IVT anti-VEGF or steroid implants (aflibercept, ranibizumab, bevacizumab, brolucizumab, pegaptanib sodium, triamcinolone, dexamethasone, fluocinolone) for more than 1 year before inclusion.
* Treatment with ocriplasmin (JETREA®) in the study eye at any time.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with eAMD with a diagnosis or under treatment for a period ≤ 1year.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Average change in best corrected visual acuity (BCVA) from baseline to month 12. | From baseline and then at each of the subsequent visits until month 12.
  BCVA will be assessed on both eyes, using best correction determined from protocol refraction. Measurements will be taken in a sitting position using ETDRS-like visual acuity testing charts at a starting distance of 4 meters.
Average change in BCVA from baseline to month 24. | From baseline and then at each of the subsequent visits until month 24.
  BCVA will be assessed on both eyes, using best correction determined from protocol refraction. Measurements will be taken in a sitting position using ETDRS-like visual acuity testing charts at a starting distance of 4 meters.

SECONDARY OUTCOMES:
Proportion of patients gaining ≥5, ≥10, ≥15 letters in BCVA at month 12. | From baseline through month 12.
  BCVA will be assessed on both eyes, using best correction determined from protocol refraction. Measurements will be taken in a sitting position using ETDRS-like visual acuity testing charts at a starting distance of 4 meters.
  The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Proportion of patients gaining ≥5, ≥10, ≥15 letters in BCVA at month 24. | From baseline through month 24.
  BCVA will be assessed on both eyes, using best correction determined from protocol refraction. Measurements will be taken in a sitting position using ETDRS-like visual acuity testing charts at a starting distance of 4 meters.
  The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Proportion of patients with BCVA ≥69 letters at month 12. | From baseline through month 12.
  BCVA will be assessed on both eyes, using best correction determined from protocol refraction. Measurements will be taken in a sitting position using ETDRS-like visual acuity testing charts at a starting distance of 4 meters.
  The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Proportion of patients with BCVA ≥69 letters at month 24. | From baseline through month 24.
  BCVA will be assessed on both eyes, using best correction determined from protocol refraction. Measurements will be taken in a sitting position using ETDRS-like visual acuity testing charts at a starting distance of 4 meters.
  The BCVA letter score ranges from 0 to 100 (best score), and a gain in BCVA from baseline indicates an improvement in visual acuity.
Average change in central retinal thickness (CRT) from baseline to month 12. | From baseline to month 12.
  Central retinal thickness refers to the measurement of the retinal tissue thickness in the central region of the retina, assessed using Optical Coherence Tomography (OCT).
Average change in CRT from baseline to month 24. | From baseline to month 24.
  Central retinal thickness refers to the measurement of the retinal tissue thickness in the central region of the retina, assessed using OCT.
Proportion of patients without fluid at foveal centre at month 12. | Month 12.
  Fluid at foveal centre is measured using OCT.
Proportion of patients without fluid at foveal centre at month 24. | Month 24.
  Fluid at foveal centre is measured using OCT.
Total number of visits during the two-year treatment period. | From baseline through end of study (24 months).
  Count of the number of visits each participant performed during the two-year treatment period.
Total number of intravitreal injections during the two-year treatment period. | From baseline through end of study (24 months).
  Count of the intravitreal injections each participant received during the two-year treatment period.
Proportion of patients with ≥ 12, ≥ 16, ≥20 weeks interval at month 12. | Month 12.
  Proportions are based on the number of participants who have not discontinued the study at the end of the study. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit.
Proportion of patients with ≥ 12, ≥ 16, ≥20 weeks interval at month 24. | Month 24.
  Proportions are based on the number of participants who have not discontinued the study at the end of the study. The treatment interval at a given visit is defined as the treatment interval decision followed at that visit.
Proportion of accurate alert flags of the OKKO-identified alerts/patient-driven alerts/clinic-identified alerts. | From baseline to the end of the study.
  Accurate alert flags are measured as similar change in clinical status of the OKKO-identified alerts/patient-driven alerts/clinic-identified alerts.
Proportion of inaccurate alert flags of the OKKO-identified alerts/patient-driven alerts/clinic-identified alerts. | From baseline to the end of the study.
  Inaccurate alert flags are measured as no correlation change in clinical status found of the OKKO-identified alerts/patient-driven alerts/clinic-identified alerts.
Adherence to the home monitoring. | From baseline to the end of the study.
  Adherence determined by patients who use the application to home-monitor VA and metamorphopsia at least weekly and have no more than 2 breaks of 3 weeks in a year.
Costs assigned to National Health System at month 12. | Month 12.
  Costs assigned to National Health System are estimated through eCRF information such as number of visits, serious adverse events (SAEs) and hospitalizations.
Costs assigned to National Health System at month 24. | Month 24.
  Costs assigned to National Health System are estimated through eCRF information such as number of visits, SAEs and hospitalizations.
Societal costs at month 12. | Month 12.
  Societal costs are assessed using a Value-based Healthcare Questionnaire, to be filled by participant and accompaniments.
Societal costs at month 24. | Month 24.
  Societal costs are assessed using a Value-based Healthcare Questionnaire, to be filled by participant and accompaniments.
Average change in National Eye Institute Visual Functioning Questionnaire 25 (NEI-VFQ-25) from baseline to month 12. | From baseline to month 12.
  NEI-VFQ-25 is a validated questionnaire used to assess vision-specific health-related quality of life. All items are scored so that a higher score represents better functioning and each item is converted to a 0 to 100 scale.
Average change in EQ-5D five-level (EQ-5D-5L) descriptive system from baseline to month 12. | From baseline to month 12.
  EQ-5D-5L is a validated questionnaire used to measure patient-reported health status and utility values. The questionnaire creates a 5-digit code from five health dimensions, scored as five levels, and the higher score represents worse outcome. The EQ-5D-5L also includes the EuroQol Visual Analogue Scale (EQ-VAS) on a 0 to 100 scale for self-rated health, which higher score means better outcome.
Average change in National Eye Institute Visual Functioning Questionnaire 25 (NEI-VFQ-25) from baseline to month 24. | From baseline to month 24.
  NEI-VFQ-25 is a validated questionnaire used to assess vision-specific health-related quality of life. All items are scored so that a higher score represents better functioning and each item is converted to a 0 to 100 scale.
Average change in EQ-5D five-level (EQ-5D-5L) descriptive system from baseline to month 24. | From baseline to month 24.
  EQ-5D-5L is a validated questionnaire used to measure patient-reported health status and utility values. The questionnaire creates a 5-digit code from five health dimensions, scored as five levels, and the higher score represents worse outcome. The EQ-5D-5L also includes the EuroQol Visual Analogue Scale (EQ-VAS) on a 0 to 100 scale for self-rated health, which higher score means better outcome.
System usability scale (SUS) score. | Month 12.
  To evaluate user satisfaction and perceived usability of the system at month 12. The SUS uses a 0 to 5 scale for each sentence, which higher scores indicate better outcomes.
Net promoter score (NPS). | Month 12.
  To evaluate user satisfaction and perceived usability of the system at month 12. The NPS uses a 0 to 10 scale, which higher score indicates better outcome.
Frequency of adverse events (AEs) at month 12. | From baseline to month 12.
  To evaluate the safety associated with the inclusion of a home monitoring app in the eAMD patient pathway with respect to AEs.
Frequency of SAEs at month 12. | From baseline to month 12.
  To evaluate the safety associated with the inclusion of a home monitoring app in the eAMD patient pathway with respect SAEs.
Frequency of AEs at month 24. | From baseline to month 24.
  To evaluate the safety associated with the inclusion of a home monitoring app in the eAMD patient pathway with respect to AEs.
Frequency of SAEs at month 24. | From baseline to month 24.
  To evaluate the safety associated with the inclusion of a home monitoring app in the eAMD patient pathway with respect to SAEs.

CONTACTS AND LOCATIONS:
Locations (8):
- Portugal (8):
  - Espaço Médico de Coimbra, Lda., Coimbra
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Unidade Local de Saúde de Leiria, E.P.E., Leiria
  - Instituto Português de Microcirurgia Ocular, Lda., Lisbon
  - Unidade Local de Saúde de Lisboa Ocidental - Hospital de Egas Moniz, Lisbon
  - Unidade Local de Saúde Loures-Odivelas, Loures
  - Unidade Local de Saúde de Santo António, E.P.E., Porto
  - Unidade Local de Saúde de São João, E.P.E., Porto